CLINICAL TRIAL: NCT04007107
Title: A Trial to Compare the Injection Site Pain Experience of 0.25 mg Semaglutide sc Administered by 2 Different Products
Brief Title: A Study Comparing the Injection Site Pain Experience After the Injection of 2 Different Solutions of Semaglutide With 2 Different Injection Pens, a Compound for the Treatment of Type 2 Diabetes and Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS-4582; 2019-002284-10 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1233-9590 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers Diabetes Mellitus, Type 2; Healthy Volunteers Overweight; Healthy Volunteers Obesity
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV3396 followed by PDS290 (Experimental): The 2 treatments will be administered at least 30 minutes apart, one in each side of the stomach
  Interventions: Drug: Semaglutide (administered by DV3396 pen); Drug: Semaglutide (administered by PDS290 pen)
- PDS290 followed by DV3396 (Experimental): The 2 treatments will be administered at least 30 minutes apart, one in each side of the stomach
  Interventions: Drug: Semaglutide (administered by DV3396 pen); Drug: Semaglutide (administered by PDS290 pen)

INTERVENTIONS:
Drug: Semaglutide (administered by DV3396 pen) — Subjects will receive 1 single dose of semaglutide 0.25 mg on 1 day
Drug: Semaglutide (administered by PDS290 pen) — Subjects will receive 1 single dose of semaglutide 0.25 mg on 1 day

SUMMARY:
This study in healthy men and women compares the injection site experience of the DV3396 pen to that of the PDS290 pens when both pens are used to deliver 0.25 mg semaglutide subcutaneously (sc, under the skin). Participants will receive 2 single doses of semaglutide 0.25 mg on 1 day. The 2 injections will be given at least 30 minutes apart, one in each side of the stomach. Participants will be in the clinic research center for 1 day. A follow-up phone call will take place between 4 and 5 weeks after the injections were given.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female subjects, aged 18 to 75 years (both inclusive) at the time of signing informed consent.
* BMI equal to or above 25.0 kg/m^2
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram, and clinical laboratory tests performed during the screening visit, as judged by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to the study product or related products.
* Previous participation in this study. Participation is defined as having received investigational product.
* Woman who is pregnant or breast-feeding or intends to become pregnant within 4 weeks after administration of the study drug, or is of childbearing potential and not using highly effective contraceptive methods with her fertile male sexual partner
* Participation in a drug study within 60 days prior to drug administration in the current study. Participation in more than 4 other drug studies in the 12 months prior to drug administration in the current study.
* Any disorder that in the Investigator's opinion might jeopardize subject's safety, evaluation of results, or compliance with the protocol.
* Glycosylated haemoglobin (HbA1c) equal to or above 6.5% at screening.
* Supine blood pressure at screening (after resting for at least 5 minutes) outside the range of 90 to 160 mmHg for systolic or 45 to 89 mmHg for diastolic.
* Supine pulse rate (as part of vital signs) (after resting for at least 5 minutes) outside the range of 40 to 100 beats per minute.
* Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication, contraceptives, and occasional use of paracetamol (paracetamol not allowed within 24 hours prior to drug administration), within 14 days prior to drug administration.
* Diagnostic test results positive for human immunodeficiency virus (HIV)-1 or HIV-2 infection.
* Diagnostic test results positive for hepatitis B or hepatitis C infection.
* Mental incapacity, language barriers, or unwillingness to comply with the requirements of the protocol, which may preclude adequate understanding or cooperation during the study as judged by the Investigator.
* Average intake of more than 21 units of alcohol per week for male subjects and more than 14 units per week for female subjects: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits.
* Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening and admission to the clinical research center.
* Use of tobacco and nicotine products, defined as any of the below:
* Smoking more than 1 cigarette or the equivalent per day on average
* Not able or willing to refrain from smoking and the use of nicotine substitute products during the in-house period
* Blood donation, plasma donation or blood draw (as declared by the subject or reported in the medical records):
* In excess of 400 mL within the past 90 days prior to the day of screening
* In excess of 50 mL within the past 30 days prior to the day of screening
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by the subject or reported in the medical records)
* Subjects with a history of malignant neoplasms within the past 5 years prior to screening.
* Presence or history of pancreatitis (acute or chronic; as declared by the subject or reported in the medical records).
* Subject is not able to understand and read English or Dutch, or subject is not able to understand and comply with the study requirements.
* Subject depends on the Sponsor, the Investigator, or the study center, or subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the study.
* Vulnerable subject (eg, person kept in detention) who may have an increased likelihood of being wronged or of incurring additional harm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Snitker S, Andersen A, Lindskov PS, van Marle S, Sode BF, Sparre T. Comparison of the injection-site experience of semaglutide in a single-dose and a multidose pen-injector. Diabetes Obes Metab. 2022 Aug;24(8):1643-1646. doi: 10.1111/dom.14718. Epub 2022 May 20. No abstract available. PMID 35434913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in the Netherlands.
Pre-assignment Details: Participants were randomised in a 2×2 scheme evenly to 4 sequences (A, B, C and D) of either DV3396 or PDS290 and side of injection (right/left) on abdomen.
Groups:
- Sequence A: DV3396 (Right) Then PDS290 (Left): Participants were to receive a subcutaneous (s.c.) injection of DV3396 product (0.25 milligrams (mg) of semaglutide) on the right side of abdomen (in treatment period 1); followed by an s.c. injection of PDS290 product (0.25 mg of semaglutide) on the left side of abdomen (in treatment period 2). The 2 products were administered on the same day (Day 1) with at least 30 minutes apart from each other.
- Sequence B: DV3396 (Left) Then PDS290 (Right): Participants were to receive an s.c. injection of DV3396 product (0.25 mg of semaglutide) on the left side of abdomen (in treatment period 1); followed by an s.c. injection of PDS290 product (0.25 mg of semaglutide) on the right side of abdomen (in treatment period 2). The 2 products were administered on the same day (Day 1) with at least 30 minutes apart from each other.
- Sequence C: PDS290 (Right) Then DV3396 (Left): Participants were to receive an s.c. injection of PDS290 product (0.25 mg of semaglutide) on the right side of abdomen (in treatment period 1); followed by an s.c. injection of DV3396 product (0.25 mg of semaglutide) on the left side of abdomen (in treatment period 2). The 2 products were administered on the same day (Day 1) with at least 30 minutes apart from each other.
- Sequence D: PDS290 (Left) Then DV3396 (Right): Participants were to receive an s.c. injection of PDS290 product (0.25 mg of semaglutide) on the left side of abdomen (in treatment period 1); followed by an s.c. injection of DV3396 product (0.25 mg of semaglutide) on the right side of abdomen (in treatment period 2). The 2 products were administered on the same day (Day 1) with at least 30 minutes apart from each other.
Period: Treatment Period 1 (Day 1)
Arm/Group | Sequence A: DV3396 (Right) Then PDS290 (Left) | Sequence B: DV3396 (Left) Then PDS290 (Right) | Sequence C: PDS290 (Right) Then DV3396 (Left) | Sequence D: PDS290 (Left) Then DV3396 (Right)
Started | 26 | 26 | 25 | 26
Full Analysis Set (FAS) | 26 | 26 | 25 | 26
Safety Analysis Set (SAS) | 26 | 26 | 25 | 26
Per Protocol (PP) Set | 26 | 25 | 25 | 26
Completed | 26 | 26 | 25 | 26
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 1)
Arm/Group | Sequence A: DV3396 (Right) Then PDS290 (Left) | Sequence B: DV3396 (Left) Then PDS290 (Right) | Sequence C: PDS290 (Right) Then DV3396 (Left) | Sequence D: PDS290 (Left) Then DV3396 (Right)
Started | 26 | 26 | 25 | 26
Completed | 26 | 25 | 25 | 26
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who had received at least 1 injection of semaglutide (included any skin contact with trial product whether the injection was completed or not).
Groups:
- Overall Study: Participants were to receive 2 s.c. injections of 0.25 mg semaglutide; 1 each of PDS290 product and DV3396 product from any of the sequences A/B/C/D on Day 1. The 2 products were administered at least 30 minutes apart from each other.
Arm/Group | Overall Study
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Black or African American | 1
  Native Hawaiian or other Pacific Islan | 0
  White | 98
  White + Black or African American | 0
  White + Asian | 2
  Asian + Black or African American | 0
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Injection Site Pain
Description: The intensity of injection site pain was measured on a visual analogue scale (VAS). The VAS consists of a horizontal 100 millimetres (mm) line where 0 mm corresponded to no pain and 100 mm corresponded to unbearable pain. After each injection, the participants rated their pain perception at the VAS by marking a vertical line across the 100 mm line. The distance (mm) between the endpoint "no pain" and the vertical line on the VAS was recorded and analysed.
Time Frame: After 1 minute of each injection (Day 1)
Population: The per protocol (PP) set included all participants who had received both injections of semaglutide and had completed both intensity of injection site pain assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DV3396: Participants were to receive a s.c. injection of DV3396 product (0.25 mg of semaglutide) on either (left or right) sides of abdomen in any of the sequences A/B/C/D on Day 1.
- PDS290: Participants were to receive a s.c. injection of PDS290 product (0.25 mg of semaglutide) on either (left or right) sides of abdomen in any of the sequences A/B/C/D on Day 1.
Arm/Group | DV3396 | PDS290
Number analyzed (Participants) | 102 | 102
score on a scale | 35.1 (23.1) | 4.4 (7.5)
Statistical Analysis 1: Comparison: DV3396 vs PDS290; The intensity of pain was analysed by a fixed analysis of variance model with VAS score as the dependent variable, and product, injection side (right side, left side), injection number (first injection, second injection), and participant as fixed effects; Test type: Other — Comparison; p < 0.0001, ANOVA; Estimated treatment difference = 30.7, 95% CI 2-sided [26.6 to 34.8]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 28. Results are based on the safety analysis set which included all participants who had received at least 1 injection of semaglutide (included any skin contact with trial product whether the injection was completed or not).
Description: All presented adverse events are treatment emergent adverse events (TEAEs). TEAE was defined as an event that had onset date on or after the day of first injection and no later than 28 days after the day of last injection. The trial was crossover and injections were given only 30 minutes apart. Therefore it was not possible to say which product the AE was related to. Hence, AE data are presented for the overall study.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 15/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=103)
Nausea (Gastrointestinal disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04007107/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT04007107/SAP_001.pdf